CLINICAL TRIAL: NCT01588548
Title: A Phase I, Open-Label, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumour Activity of Ascending Doses of AZD1208 in Patients With Advanced Solid Malignancies Including Malignant Lymphoma
Brief Title: Global Phase1 Study to Assess the Safety and Tolerability of AZD1208 in Advanced Solid Tumors and Malignant Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4510C00005
Record Dates: First submitted 2012-04-27; First posted 2012-05-01 (Estimated); Results first posted 2015-08-19 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-10

CONDITIONS: Advanced Solid Malignancies; Malignant Lymphoma
Keywords: Advanced solid malignancies; Malignant lymphoma
MeSH Terms: conditions — Lymphoma | interventions — AZD1208

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AZD1208 (Active Comparator)
  Interventions: Drug: AZD1208

INTERVENTIONS:
Drug: AZD1208 — Dose of AZD1208 will be escalated from 120mg to a maximum tolerated dose

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of AZD 1208 up to a maximum tolerated dose (MTD) and define the dose(s) for further clinical evaluation when given daily to patients with advanced solid malignancies including malignant lymphoma

DETAILED DESCRIPTION:
A Phase I, Open-Label, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumour Activity of Ascending Doses of AZD1208 in Patients with Advanced Solid Malignancies including Malignant Lymphoma

ELIGIBILITY:
Inclusion Criteria:

* Patients who have signed this Written Informed Consent Form after a full explanation about the participation in this study
* Patients aged 18 years or older Patients diagnosed with a solid malignant tumour or malignant lymphoma that is refractory to standard therapies or for which no standard therapies exist
* Patients with good physical conditions (you can walk and can look after yourself) within the last 2 weeks.
* Patients who have at least one lesion that can be accurately assessed

Exclusion Criteria:

* Patients who have recently received or are receiving prohibited medications or treatments
* Patients who have any unresolved side effects of previous treatments
* Patients who have spinal cord compression or brain metastases
* Patients who have severe systemic diseases (e.g., uncontrolled hypertension, hepatitis B, hepatitis C and human immunodeficiency virus [HIV] infection)
* Patients with significant abnormal ECG findings

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Neumann, MSD, Study Director — AZ
Locations (3):
- Research Site, Chūōku, Japan
- United Kingdom (2):
  - Research Site, Manchester
  - Research Site, Surrey

REFERENCES:
- See also: CSR_Synopsis_D4510C00005.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=457&filename=CSR_Synopsis_D4510C00005.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 43 patients were enrolled to the study, of which 35 recieved doses of AZD1208 between 120mg and 800mg. The other 8 patients did not receive AZD1208.
Groups:
- AZD1208 120mg; AZD1208 240mg; AZD1208 360mg; AZD1208 540mg; AZD1208 700mg; AZD1208 800mg: Once daily continuous dosing schedule.
Period: Overall Study
Arm/Group | AZD1208 120mg | AZD1208 240mg | AZD1208 360mg | AZD1208 540mg | AZD1208 700mg | AZD1208 800mg
Started | 3 | 7 | 6 | 7 | 6 | 6
Cycle 1 Day 21 | 3 | 5 | 2 | 5 | 3 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 7 | 6 | 7 | 6 | 6
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 1 | 2 | 3
Not completed — Adverse Event | 0 | 0 | 1 | 2 | 1 | 0
Not completed — Condition Under Investigation Worsened | 3 | 6 | 4 | 4 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD1208 120mg | AZD1208 240mg | AZD1208 360mg | AZD1208 540mg | AZD1208 700mg | AZD1208 800mg | Total
Number analyzed (Participants) | 3 | 7 | 6 | 7 | 6 | 6 | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.0 (9.00) | 59.4 (9.81) | 63.5 (14.38) | 62.3 (17.01) | 66.5 (12.85) | 60.8 (12.45) | 61.7 (12.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 2 | 3 | 4 | 3 | 18
  Male | 1 | 3 | 4 | 4 | 2 | 3 | 17

OUTCOME MEASURES:

1. Primary Outcome: Best Objective Response Based on RECIST Criteria (Evaluable for Response Analysis Set for RECIST Criteria)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), disappearance of all target lesions (TL)s since baseline and any pathological lymph nodes selected as TLs must have a reduction in short axis to <10 mm; Partial Response (PR), at least a 30% decrease in the sum of diameters of TLs; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD; Progressive Disease (PD), at least a 20% increase in the sum of diameters of TLs and an absolute increase of at least 5 mm; Not Evaluable (NE), this is only relevant if any of the TLs were not assessed or not evaluable or had a lesion intervention at this visit, also note that if the sum of diameters meets the progressive disease criteria, progressive disease overrides not evaluable as a TL response. Best objective response is the best response a patient experiences over the randomised treatment period.
Time Frame: Measurements occur at screening (<=28 days before start of study treatment), every 6 weeks (+/-1 week) up to 12 weeks and then every 12 weeks (+/-1 week) until discontinuation of study treatment or withdrawal of consent, starting from Day 1 of Cycle 1
Population: All patients who were evaluable for Response analysis set for RECIST criteria
Measure: Number; unit: Participants
Arm/Group | AZD1208 120mg | AZD1208 240mg | AZD1208 360mg | AZD1208 540mg | AZD1208 700mg | AZD1208 800mg
Number analyzed (Participants) | 3 | 7 | 5 | 7 | 6 | 5
Participants
  CR | 0 | 0 | 0 | 0 | 0 | 0
  PR | 0 | 0 | 0 | 0 | 0 | 0
  SD >=6 weeks (unconfirmed CR or PR) | 0 | 0 | 0 | 0 | 0 | 0
  SD >=6 weeks (SD) | 2 | 5 | 1 | 3 | 1 | 1
  PD (RECIST progression) | 1 | 2 | 3 | 3 | 2 | 3
  PD (Death) | 0 | 0 | 0 | 0 | 1 | 0
  Not evaluable (SD < 6 weeks) | 0 | 0 | 1 | 0 | 2 | 0
  Not evaluable(Incomplete postbaseline assessments) | 0 | 0 | 0 | 1 | 0 | 1

ADVERSE EVENTS:
Arm/Group | AZD1208 120mg | AZD1208 240mg | AZD1208 360mg | AZD1208 540mg | AZD1208 700mg | AZD1208 800mg
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/7 | 2/6 | 2/7 | 2/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 6/6 | 7/7 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD1208 120mg (N=3) | AZD1208 240mg (N=7) | AZD1208 360mg (N=6) | AZD1208 540mg (N=7) | AZD1208 700mg (N=6) | AZD1208 800mg (N=6)
Bacterial Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Balance Disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
General Physical Health Deterioration (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD1208 120mg (N=3) | AZD1208 240mg (N=7) | AZD1208 360mg (N=6) | AZD1208 540mg (N=7) | AZD1208 700mg (N=6) | AZD1208 800mg (N=6)
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 0
Oral Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Bacterial Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Lung Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Vaginal Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 4 | 2 | 4 | 3 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 3 | 2 | 4 | 2 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 1 | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 4 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 2 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Balance Disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Disturbance In Attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neuropathy Peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sensory Disturbance (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dry Eye (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dysaesthesia Pharynx (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 5 | 5 | 6 | 5 | 6
Nausea (Gastrointestinal disorders) | 1 | 6 | 3 | 7 | 5 | 4
Vomiting (Gastrointestinal disorders) | 0 | 6 | 1 | 5 | 4 | 3
Abdominal Pain (Gastrointestinal disorders) | 0 | 3 | 2 | 2 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 2 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 0
Hepatic Pain (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal Tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 2 | 1 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0
Rash Macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Nail Disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Skin Fissures (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Skin Mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 3 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0
Cystitis Noninfective (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pelvic Pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 3 | 3 | 4 | 5
Pyrexia (General disorders) | 0 | 1 | 3 | 0 | 2 | 0
Chest Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Device Occlusion (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
General Physical Health Deterioration (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hernia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Mucosal Inflammation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Suprapubic Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Platelet Count Decreased (Investigations) | 2 | 2 | 1 | 2 | 1 | 1
White Blood Cell Count Decreased (Investigations) | 2 | 3 | 1 | 2 | 1 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 2 | 1 | 2 | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 2 | 0 | 1 | 0 | 0
Blood Creatinine Increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 1
Lymphocyte Count Decreased (Investigations) | 0 | 1 | 2 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0
Neutrophil Count Decreased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0
Oxygen Saturation Decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood Urea Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Breath Sounds Abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram Qt Prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal Stoma Output Decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Weight Decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Arthropod Bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AstraZeneca will manage the publication of the results of the Clinical Trial in partnership with the authors. AstraZeneca recognises that Institutions/Investigators may wish to make publications regarding Clinical Trial results. The Institution/Investigator agrees to collaborate in good faith with AstraZeneca. Prior to any such publication, the Institution/Investigator shall provide AstraZeneca with preliminary data and drafts of proposed publications.